CLINICAL TRIAL: NCT02708979
Title: StrEat - Stress and Eating Behavior
Brief Title: Stress and Eating Behavior Among University Students - an Randomized Controlled Trial
Acronym: StrEat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anders M Sjödin, MD, PhD, Professor, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: B321
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Stress
Keywords: Stress; Eating

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- University Exam Period (Active Comparator): This visit takes place the week before an exam at the university assuming that this will induce a stress response. Measurements (see description elsewhere) are being taken within 1-2 weeks prior to an university exam.
  Interventions: Other: University exam-period
- University Non-exam Period (Placebo Comparator): This visit takes place several weeks post and prior to an exam at the university assuming that students will not be stressed in this period. Measurements (see description elsewhere) are being taken in a control-period without exams (at least 4 weeks after and 4 weeks prior to an exam)
  Interventions: Other: University non-exam-period

INTERVENTIONS:
Other: University exam-period — This visit takes place one week prior to an exam at the university assuming that students will be stressed in this period.
  Arms: University Exam Period
Other: University non-exam-period — This visit takes place several weeks post and prior to an exam at the university assuming that students will not be stressed in this period.
  Arms: University Non-exam Period

SUMMARY:
The high worldwide prevalence of overweight and obesity as well as metabolic and disease consequences, are well-documented. The positive energy balance underlying obesity is attributable to excess energy intake and/or insufficient energy expenditure. However, it seems that the increase in mean body weight can be sufficiently explained by increases in mean energy intake. It has been proposed that this overeating is partly caused by increased availability of highly processed energy dense, high reward foods. Psychosocial stress and sleep insufficiency is pervasive in industrialized societies. A growing body of evidence suggests stress to be involved in obesity, although it is unknown whether stress is a cause or consequence. Stress affecting dietary intake; skewing intake towards greater consumption of highly palatable energy dense foods, also referred to as high reward foods. A causal relationship between stress and reward seeking behavior is supported by findings from animal studies reporting rewarding behavior by consumption of sweet tasting food in response to a stressor.

Our aim is to investigate differences in purchases of particular food-items in free living individuals, during a stressful (upcoming exam) and non-stressful (no upcoming exam) period.

Hypothesis: Participants will purchase more high reward foods during the pre-exam period, compared to the control non-exam period.

DETAILED DESCRIPTION:
STUDY METHODS

Study design:

The study is a randomized controlled two-armed cross-over intervention study. The study is carried out in 50 healthy university students, both genders. In random order the participants will be investigated during stressful-period (prior to an exam) and a non-stressful (control period) period. Each participant will take part in all together four visits, two in the stressful period and two visits in the non-stressful period.

The study will take place, at the Department of Nutrition, Exercise and Sports (NEXS), Faculty of Science at the University of Copenhagen, Rolighedsvej 26, 1958 Frederiksberg C. Recruitment will take place at the University of Copenhagen

STATISTICAL ANALYSES Analysis of the primary outcome (food choices) will be based on an ANCOVA-type linear mixed model with the intervention and allocation order as the fixed effect and person as the random effect. Analysis will be performed using the software R, SAS, STATA or SPSS. Analyses, data processing and writing of the article are expected to extend over the study period and a year beyond.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, weight stabile (defined as no weight gain/loss >3 kg during the past three months) students at the University of Copenhagen
* Age > 18 years, men and women

Exclusion Criteria:

* Purposefully seeking to lose or gain weight
* Diabetes.
* Blood donation < 1 week prior to the study and during the study
* Lactation, Pregnancy or planning of pregnancy during the study
* Inability, physically or mentally, to comply with the procedures required by the study- protocol, as evaluated by the investigator
* Participation in other clinical trials during the study
* Diagnosed with stress
* Daily use of medication influencing biomarkers of stress

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Differences in purchase of high reward foods from the gift certificates between the exam-period and non-exam period. | The outcome is assessed twice, once in the exam period (one week prior to an exam) and once in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The classification will be done blinded for the outcome assessor.

SECONDARY OUTCOMES:
Differences in Heart Rate Variability (HRV) based on a one minute breathing test between the exam-period and non-exam period. | The outcome is assessed twice, once in the exam period (one week prior to an exam) and once in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The classification will be done blinded for the outcome assessor.
Differences in morning cortisol measured in saliva between the exam-period and non-exam period. | The outcome is assessed twice, once in the exam period (one week prior to an exam) and once in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The classification will be done blinded for the outcome assessor.
Differences in insulin resistance measured by homeostatic model assessment (HOMA-IR) calculated from insulin and glucose measured in plasma between the exam-period and non-exam period. | The outcome is assessed twice, once in the exam period (one week prior to an exam) and once in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The analyses will be done blinded for the outcome assessor.
Differences in Perceived Stress (Perceived Stress Scale, PSS) between the exam-period and non-exam period. | The outcome is assessed twice, once in the exam period (one week prior to an exam) and once in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The analyses will be done blinded for the outcome assessor.
Differences in eating behavior using the "Three factor eating questionnaire" between the exam-period and non-exam period. | The outcome is assessed twice, once in the exam period (one week prior to an exam) and once in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The analyses will be done blinded for the outcome assessor.
Differences in sleep habits using the "Pittsburgh sleep quality index" between the exam-period and non-exam period. | The outcome is assessed twice, once in the exam period (one week prior to an exam) and once in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The analyses will be done blinded for the outcome assessor.
Differences in sleep duration measured by ActiGraph between the exam-period and non-exam period. | The outcome is assessed twice, in the exam period (one week prior to an exam) and in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The analyses will be done blinded for the outcome assessor.
Differences in activity measured by ActiGraph between the exam-period and non-exam period. | The outcome is assessed twice,in the exam period (one week prior to an exam) and in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The analyses will be done blinded for the outcome assessor.
Differences in blood pressure between the exam-period and non-exam period. | The outcome is assessed twice, once in the exam period (one week prior to an exam) and once in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The analyses will be done blinded for the outcome assessor.
Differences in Perceived Stress ( questionaire: RESTQ-76 sport) between the exam-period and non-exam period. | The outcome is assessed twice, once in the exam period (one week prior to an exam) and once in the non-exam period (four to five weeks prior and post an exam ) Data are analyzed after last subject last visit (May 2016)
  The analyses will be done blinded for the outcome assessor.

CONTACTS AND LOCATIONS:
Overall Officials: Anders M Sjödin, PhD, Study Chair — University of Copenhagen, NEXS; Mads F Hjorth, PhD, Principal Investigator — University of Copenhagen; Julie B Schmidt, PhD, Principal Investigator — University of Copenhagen, NEXS
Locations (1):
- Nutrition, Exercise and Sports, Frederiksberg, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No